CLINICAL TRIAL: NCT00465400
Title: Quantification of Oxidative Stress in Patients With Age-Related Macular Degeneration Prior to and After Photodynamic Therapy: a Comet Assay Analysis
Brief Title: Oxidative Stress in Patients With Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Selim Orgul, University Hospital, Basel, Switzerland
Other Study IDs: 086-Mom-2006-004
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Macular Degeneration
Keywords: exudative age-related macular degeneration (AMD); non-exudative age-related macular degeneration (AMD); oxidative stress; photodynamic therapy
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
First, to quantify, by means of comet assay analysis, systemic oxidative stress in patients with non-exudative and exudative age-related macular degeneration (AMD) and compare results to healthy controls.

Second, to quantify systemic oxidative stress in patients with exudative AMD prior to and after photodynamic (PDT) therapy.

DETAILED DESCRIPTION:
Oxidative stress is the major factor that plays a role in the pathogenesis of age-related macular degeneration (AMD), which is a leading cause of blind registration in the developed world. The term oxidative stress refers to reversible damage to molecules, such as for example DNA, by reactive forms of oxygen (eg. free oxygen radicals). This damage is repaired is normally repaired in our body.

AMD is classified in two forms: the dry (non-exudative) and wet (exudative) form. The exudative form of AMD occurs when new blood vessels form to improve the blood supply to retinal tissue. However, the new blood vessels are very delicate and break easily, causing bleeding and serious vision loss. The standardized method used to treat exudative AMD is photodynamic therapy (PDT). This treatment is based upon the infusion of a drug that can be activated by light and produces free radicals that destroy these newly formed vessels. In other words, these new vessels are destroyed by an iatrogenic source of oxidative stress. This means that the factor that originally caused the disease AMD, namely oxidative stress, is finally used as a form of treatment- to destroy these newly formed blood vessels.

In the present study we would like to quantify in a first step the level of systemic oxidative stress in patients with non-exudative and exudative AMD and compare to healthy controls. In a second step we would like to test whether the treatment (PDT) for patients with exudative AMD additionally increases systemic oxidative stress. Oxidative stress is quantified in our laboratory by means of single cell gel electrophoresis or comet assay.

ELIGIBILITY:
Inclusion Criteria:

For patients with dry non- exudative AMD:

* Patients between the ages of 50 and 85 yr inclusive.
* Study eye must have a diagnosis of nonexudative "dry" AMD with ≥10 large soft, semisoft, and/or confluent drusen within 3,000 nm of the foveal center.
* Study eye must have a best corrected visual acuity using the ETDRS chart between 0.1 patem and 0.8 patem inclusive.
* Geographic atrophy is allowed as long as it is less than 3 disc diameters within 3,000 nm of the foveal center.
* Study eye must not have conditions that limit the view of the fundus.

For patients with exudative AMD with clinical indication for PDT treatment:

* Patients between the ages of 50 and 85 yrs with exudative AMD with clinical indication for PDT treatment.
* Primary or recurrent subfoveal CNV due to AMD
* Central 1-mm retinal thickness (optical coherence tomography) > 300 um
* Best-corrected visual acuity, using ETDRS charts, of > 0.05patem
* Evidence of recent disease progression, including the loss of at least 1 line of visual acuity or macular hemorrhage within the previous 12 wks.

For healthy subjects:

* An intraocular pressure < 20 mmHg
* Normal blood pressure (100-140/60-90mm Hg)
* Best corrected visual acuity, using EDTRS charts of above 0.6 patem in both eyes
* No pathological findings upon slit-lamp examination and indirect fundoscopy

Exclusion Criteria:

* History of other ocular or systemic disease
* History of chronic or current systemic or topical medication, or of significant drug or alcohol abuse(significant is defined as that which may influence results of the study
* History of ocular trauma or intraocular surgery within the past 6 months
* History of infection or inflammation within the past 3 months

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgül, MD, Study Director — University Eye Clinic Basel
Locations (1):
- University Eye Clinic Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Mayne ST. Antioxidant nutrients and chronic disease: use of biomarkers of exposure and oxidative stress status in epidemiologic research. J Nutr. 2003 Mar;133 Suppl 3:933S-940S. doi: 10.1093/jn/133.3.933S. PMID 12612179